CLINICAL TRIAL: NCT04610801
Title: A Randomized Placebo Control Trial to Evaluate the Efficacy of Xylitol Nasal Spray vs. Placebo for Acute COVID-19 Infection
Brief Title: Evaluation of the Efficacy of Xylitol Nasal Spray Against SARS-CoV-2
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Period Ended/ Not Completed
Sponsor: Larkin Community Hospital (Other)
Collaborators: Ferrer Medical Innovations (Unknown); Xlear, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: LCH-3-082020
Record Dates: First submitted 2020-10-26; First posted 2020-11-02 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Covid19
Keywords: Covid 19; Intranasal Spray; Therapeutics
MeSH Terms: conditions — COVID-19 | interventions — Nasal Sprays; xylitol and grapefruit seed extract drug combination

STUDY DESIGN:
Who Masked: Care Provider
Masking Description: Masking to care providers
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- No treatment (No Intervention): No treatment given
- Treatment (Experimental): Xylitol plus Grapefruit Seed Extract (Xlear) nasal spray, 2 puffs per nosetrils, every 6 hours
  Interventions: Drug: Nasal Spray
- Placebo (Placebo Comparator): Saline nasal spray, 2 puffs per nosetrils, every 6 hours
  Interventions: Drug: Nasal Spray

INTERVENTIONS:
Drug: Nasal Spray — Randomized to placebo and Xlear
  Other Names: Xlear
  Arms: Placebo; Treatment

SUMMARY:
The purpose of this study is to assess the efficacy of Xylitol plus Grapefruit Seed Extract (Xlear) nasal spray as an adjunct treatment of COVID-19.

DETAILED DESCRIPTION:
After being informed about the study and potential risk, all patients giving written informed consent will undergo a brief screening period to determine eligibility for the study. Once eligibility is confirmed, patients who meet the eligibility requirements will be randomized placebo control manner. Patient will be assigned to Xlear (2 puffs per nosetrils, every 3-4 hours a day) or placebo. Patient will be followed for 1 week. Inflammatory markers will be obtained on Day 4 and repeat COVID-19 RT PCR on Day 7. Follow up will be done on Day 14 for all patients.

ELIGIBILITY:
Inclusion Criteria:

1. Adults of ages 18 to 90 years of both sexes
2. With positive SARS-CoV-2 carriage confirmed by nasopharyngeal PCR
3. Signed informed consent
4. 1- Mild symptoms: Minimum respiratory symptoms or asymptomatic plus positive test
5. 2- Moderate symptoms: Respiratory symptoms such as cough, mild shortness of breath with mild oxygen desaturation(room air SpO2 <92% and >88% or <88% corrected to >92% with 2lt of oxygen)

Exclusion Criteria:

1. Patient with very low viral load (threshold cycle [Ct] > 25 per PCR).
2. Known hypersensitivity to one of the constituents, particularly to xylitol or GSE
3. Under 18 years of age
4. Women of childbearing age who are pregnant, breastfeeding mothers, and intend to become pregnant during the study period; unwilling/unable to take a pregnancy test.
5. Unable to provide informed consent or decline to consent or unwillingness to adhere to the Standard of Care protocol.
6. Patients with severe symptoms -Hypoxia (SpO2 <88% not corrected by 2 liter non-concentrated oxygen) plus severe shortness of breath
7. History of immunodeficiency or are currently receiving immunosuppressive therapy.
8. Have had a planned surgical procedure within the past 12 weeks.
9. Already part of this trial, recruited at a different hospital.
10. Patient unable to perform oro-nasopharyngeal decolonization
11. Patients with acute exacerbation of severe comorbidities like heart disorders Chronic Obstructive Pulmonary Disease (COPD), Heart Failure New York Heart Association (NYHA) Class 3 and 4 and/or diseases with severe oxygenation problems
12. Patients on Remdesivir and/or other clinical trials.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-08 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-08-08 (Actual)

PRIMARY OUTCOMES:
Change from baseline reactive to non-reactive on COVID 19 RT PCR in 7 days | Baseline and 7 days
  The COVID 19 RT PCR is the gold standard in detecting presence of COVID-19 in patients. The average time from reactivity to non-reactivity is 14 days,

SECONDARY OUTCOMES:
Change of time to clinical recovery from baseline within 7 days | Baseline and 7 days
  Change in clinical symptoms including but not limited to agnosmia, ageusia, fever, congestion and other clinical symptoms associated with mild COVID-19 infection.

CONTACTS AND LOCATIONS:
Overall Officials: Gustavo Ferrer, MD, Principal Investigator — Larkin Community Hospital
Locations (2):
- United States (2):
  - Larkin Community Hospital Palm Springs Campus, Miami, Florida
  - Larkin Community Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: No